CLINICAL TRIAL: NCT01488266
Title: Comparison of Aripiprazole Augmentation vs Switching to Different Class of Antidepressants for Patients With MDD Who Are Partially/Minimally Responsive to Current Antidepressants:Randomized, Rater-blinded, Prospective Study
Brief Title: Aripiprazole Augmentation Versus Switching to Different Class of Antidepressants in Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Korea University (Other)
Collaborators: Korea OIAA (Unknown); Taiwan Otsuka Pharm. Co., Ltd (Industry)
Responsible Party: Principal Investigator, Chansu Han, MD, PhD, MHS, Associate Professor of Psychiatry, Korea University School of Medicine, Korea University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CASCADE
Record Dates: First submitted 2011-12-04; First posted 2011-12-08 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Major Depressive Disorder
Keywords: depression; depressive; major; aripiprazole; switching; augmentation; antidepressant
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Aripiprazole; Escitalopram; Fluoxetine; Paroxetine; Sertraline; Mirtazapine; Venlafaxine Hydrochloride; Milnacipran; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- aripiprazole augmentation (Experimental)
  Interventions: Drug: Aripiprazole
- different class of antidepressant (Active Comparator)
  Interventions: Drug: switching to different class of antidepressant

INTERVENTIONS:
Drug: Aripiprazole — patients who are randomly assigned to adjunctive aripiprazole are treated with a starting dose of 2.5 (or 5) mg/day of aripiprazole, which can be increased weekly in 2.5~5mg/day increments to a maximum dose of 15 mg/day based on assessment of tolerability and clinical response. Doses can be decreased at any visit, based on tolerability; They continue to receive the same fixed-dose of the previously used antidepressant throughout the study period when patient is assigned to aripiprazole augmentation group.
  Other Names: abilify
  Arms: aripiprazole augmentation
Drug: switching to different class of antidepressant — Patients randomly assigned to switching to different antidepressant have to discontinue the previously used antidepressant and receive different antidepressant within flexible therapeutic doses as indication label information (as based on clinicians' preference and experience). Dose increase is permitted until the first 2 weeks of the study.
  Other Names: escitalopram; fluoxetine; paroxetine; sertraline; bupropion XL; mirtazapine; venlafaxine; milnacipran; duloxetine
  Arms: different class of antidepressant

SUMMARY:
The objective of this study is to compare the efficacy and safety of aripiprazole as adjunctive therapy versus switching to different class of antidepressants for treating major depressive disorder partially or minimally responsive to ongoing antidepressant treatment.

DETAILED DESCRIPTION:
Most guidelines have suggested that those nonresponders or partial responders should be considered for a switch, combination or augmentation of treatment. Traditional augmentation agents, lithium, triiodothyronine (T3), buspirone, dopamine agonists, and stimulants have been commonly used for this patient population with limited supporting data. Recently, augmentation of atypical antipsychotics with antidepressant therapy has become a more commonly accepted treatment practice. This strategy has proven to be useful for enhancement of antidepressant effect, showing increased remission rates and early treatment effects on core depressive symptoms, and comorbid symptoms as well as antidepressant- mediated side effects (e.g., sexual dysfunction). Although, we have some limited treatment options to treat such patients as described above, it is not clear which treatment option would be best or acceptable for those patients in clinical practice yet.

Among above augmentation agents, aripiprazole is the first drug approved by U.S. FDA. as an augmentation therapy to antidepressants in the treatment of patients with MDD showing imminent efficacy and reliable safety profile through adequately-powered well-designed controlled clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are older than 20 years of age have a diagnosis of MDD without psychotic features, as defined by DSM-IV-TR.
* Patients have to report an inadequate response to a current antidepressant treatment. Inadequate response to antidepressant is defined as: total score of HDRS-17 is more than 14), despite adequate dose of current antidepressant treatment for at least 6 weeks in the current episode(co-administered with ATRQ)
* Classification of antidepressants which can be included in the study(list for suggestion): Escitalopram 10~20mg/day, fluoxetine 20~40mg/day,paroxetine controlled release(CR) 25~62.5mg or paroxetine 20~40mg, sertraline 100~150mg,bupropion XL(SR) 150~300mg, mirtazapine 15~45mg,venlafaxine immediate or extended release(IR or ER) 112.5~225mg/day, duloxetine 60mg [same criteria for generic medications as brand drugs]

Exclusion Criteria:

* Those who are first episode, drug naive MDD subjects
* Those who have a current Axis I diagnosis of delirium, dementia, amnestic or other cognitive disorder, schizophrenia or other psychotic disorder, bipolar 1 or 2 disorder, eating disorder, obsessive-compulsive disorder, panic disorder, or posttraumatic stress disorder
* Those who have a clinically significant current Axis 2 diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal, or histrionic personality disorder
* Those who experience hallucinations, delusion, or any psychotic symptomatology in the current depressive episode
* Those who have met DSM-IV-TR criteria for any significant substance use disorder within the past 12 months (except nicotine)
* Those who have known allergy,hypersensitivity or previous unresponsiveness to aripiprazole or known intolerance to other study medications
* Those who have had cognitive-behavioral therapy or other psychotherapy, or they have the potential need to be treated with them during the study periods
* Those who are complicated with serious medical problem, such as severe renal, hepatic dysfunction, cardiovascular, lung, gastrointestinal, endocrine, nervous, infectious disease, or neoblastic, metabolic disease
* Those who have shown previous unresponsiveness to adequate antidepressant trials more than 2 episodes or with 3 or more antidepressant treatments
* Those who have chronic liver or renal disease
* Those who are pregnant or brest-feeding
* Those who have participated in a clinical trial with aripiprazole or any other investigational product within the past month(include randomized, double-blind, placebo-controlled or open-label study; but chart review,observational study can be enrolled)
* Those who had a history of thyroid pathology, neuroleptic malignant syndrome, or serotonin syndrome
* Those who have received adjunctive antipsychotic plus antidepressant for more than 3 weeks during the current episode
* Those who have received electroconvulsive therapy for the current episode
* Those who have shown an inadequate response to previous ECT in any episode
* Those who have a suicidal risk
* Those who are likely to require prohibited concomitant therapy during the trial
* Those who have received treatment with a monoamine oxidase inhibitor within 2 weeks prior to enrollment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-01 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Change of total score of MADRS | From baseline to end of treatment
  MADRS: montgomery Asberg Depression Rating Scale
Response rate | at 2 weeks
  response rate is defined as a reduction in MADRS total score of at least 50% relative to the beginning of the randomized phase (baseline)

SECONDARY OUTCOMES:
Response rate | at week 2,4 and 6
Remission rate | at week 2,4and 6
  remission rate is defined as an absolute MADRS total score of ≤10 at the end of treatment
Change of total score of HDRS-17 | from baseline to end of treatment
  HDRS-17: Hamilton Depression Rating Scale-17 item
Change of total score of CGI-S | from baseline to end of treatment
  CGI-S: Clinical Global Impression-Severity Score
Change of total score of IFS | from baseline to end of treatment
  IFS: Iowa Fatigue Scale
Change of total score of SDS | from baseline to end of treatment
  SDS: Sheehan Disability Scale
Patients' ratio who have have scored 1 or 2 in the score of CGI-Improvement | at the end of treatment
  CGI-I: Clinical Global Impression-Improvement Score

CONTACTS AND LOCATIONS:
Overall Officials: Changsu Han, MD,PhD, MHS, Study Chair — Korea Univ Ansan Hospital
Locations (2):
- Korean Univ Ansan Hospital; Bucheon St.Mary Hospital; DonggukUniv Gyeongju Hospital; Catholic University of Korea St. Paul's Hospital, Seoul, South Korea
- Chang Gung Memorial Hospital; Kaohsiung Medical University Chung-ho Memorial Hospital, Taipei, Taiwan